CLINICAL TRIAL: NCT07355686
Title: Success of Endodontic Regenerative Approaches in Anterior and Posterior Immature Non Vital Teeth A Randomized Controlled Clinical Trial
Brief Title: Success of Endodontic Regenerative Approaches in Anterior and Posterior Immature Non Vital Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Kholoud Emam, Teaching Assistant, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FADASU-Rec D032121
Record Dates: First submitted 2025-12-02; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Regenerative Endodontic Procedures
Keywords: regereration; immature teeth

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immature non-vital anterior teeth treated using palette rich fibrin (Active Comparator)
  Interventions: Procedure: endodontic regenerative procedure using platelet rich fibrin
- Immature non-vital anterior teeth treated using blood clot (Active Comparator)
  Interventions: Procedure: endodontic regenerative procedure using blood clot
- Immature non-vital molar teeth treated using palette rich fibrin (Active Comparator)
  Interventions: Procedure: endodontic regenerative procedure using platelet rich fibrin
- Immature non-vital molar teeth treated using blood clot (Active Comparator)
  Interventions: Procedure: endodontic regenerative procedure using blood clot

INTERVENTIONS:
Procedure: endodontic regenerative procedure using blood clot — regenerative endodontic procedure according to the American association of endodontics while using blood clot as a scaffold
  Arms: Immature non-vital anterior teeth treated using blood clot; Immature non-vital molar teeth treated using blood clot
Procedure: endodontic regenerative procedure using platelet rich fibrin — regenerative endodontic procedure according to the American association of endodontics guidelines while using Palette rich fibrin as a scaffold
  Arms: Immature non-vital anterior teeth treated using palette rich fibrin; Immature non-vital molar teeth treated using palette rich fibrin

SUMMARY:
Aim of the Study

To compare between anterior and posterior immature non vital teeth regarding:

1. Primary outcome: Resolution of apical periodontitis.
2. Secondary outcome: a) Increase in root length b) Increase in root width c) Decrease in apical area

Using the following techniques:

1. Blood clot revascularization (BC).
2. Platelet-rich fibrin (PRF).

Methods:

1. Diagnosis:

   Diagnostic data was collected & recorded in a medical & dental history sheet. A full history of the chief complaint was recorded including the intensity, nature, quality, onset, location, duration, course as well as initiating & relieving factors of pain (if present).

   Clinical Examination:
   * Visual examination using mirror & probe to detect caries, previous restorations or discoloration. - Examination of the Intraoral tissues for the detection of any swelling or sinus tract related to the tooth.
   * Palpation, Percussion, Bite & Mobility tests was done to evaluate the periapical & periodontal status of the involved tooth.
   * Periodontal probing of pocket depth was recorded for each of the involved teeth at 6 points: Mesiobuccally, Mid buccally, Distobuccally, Mesiolingually, Mid lingually & Distolingually.
   * Pulp Sensibility tests, both Thermal (cold) & Electrical was done & recorded for the involved tooth as well as the contralateral tooth, in order to affirm the diagnosis as well as to serve as a reference for follow up.

   Radiographic examination:
   * An Intraoral periapical digital radiograph with standardized paralleling angle technique using XCP film holder & standardized exposure settings (60 kV, 7 mA & 0.160) was taken pre-operatively for the involved tooth using a size 2 PSP imaging plate.
   * Pre-operative CBCT with a limited field of view (40×40) was done in which the lesion size, bone density in the area of periapical lesion & normal adjoining bony regions, & the length & width of the roots along with the diameter of the apex will be measured.
2. clinical procedure:

The clinical procedures was done (according to the guide lines of the American Association of Endodontics over 2 visits that are 2 weeks apart, unless persistence of clinical signs & symptoms occur.

First appointment:

1. Patients was given local anesthesia.
2. Dental dam isolation then access was done.
3. Minimal circumferential filing using hand files along with Copious, gentle irrigation will be done in the canals with 1.5% sodium hypochlorite ( NaOCl) (20mL) using needle with closed end and side-vents to minimize the possibility of extrusion of solutions into the periapical space and then will be irrigated with 17% ethylene diamine tetra acetic acid (EDTA) (20 mL), with irrigating needle positioned about 1 mm from root end.
4. Canals was dried using paper points.
5. Calcium hydroxide (CH) was injected using 29gauge NaviTip to the full length of the canals.
6. Access was sealed with 3-4mm of glass ionomer then patient will be dismissed for 1-4 weeks.

Second appointment: (regeneration procedure):

2 weeks after the first visit: For the four groups final visit was scheduled when tooth is asymptomatic and no signs of discharge. In cases of persistent infection one or more visits will be scheduled for discharge and disinfection.

1. The patients was given anesthesia without vasoconstrictor, proper isolation will be done; the temporary restoration and cotton pellet was removed.
2. Canals were irrigated with 20 ml of 17% EDTA for 1 minute.
3. Canals were then dried using sterile paper points.
4. In group I and group III: sterile hand file size #50 will be used in sharp strokes 2mm beyond the apex into the peri-apical tissues until bleeding is evident in cervical portion of the canal.
5. In group II and group IV: The prepared PRF will be inserted into the root canal orifice and plugged into the premeasured length of the root canal using endodontic pluggers up to 1 mm below the root canal orifice.
6. Collagen matrix was placed at the orifice, over the blood clot and white mineral trioxide aggregate (MTA )to seal the canal orifice with a wet sterile cotton pellet above. Temporary filling will be used to seal the cavity.
7. After 2 days adhesive composite resin was used to seal the access cavity.

ELIGIBILITY:
Inclusion Criteria:

* • Age 8-15.

  * Medically free.
  * Single rooted immature necrotic permanent teeth.
  * Tooth without vertical root fracture or resorption.
  * Compliant patient/parent.
  * Patient not allergic to medicaments and antibiotics necessary to complete procedure.

Exclusion Criteria:

* Avulsed teeth immediately after replantation (as revitalization may occur naturally).
* Luxation injuries.
* Impossibility of adequate tooth isolation.
* Teeth with extensive loss of coronal tissue that require restoration with a post that will occupy the space required for blood clot formation.
* Medically compromised patients.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-09-02 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
percent of change in apical lesion size | 1 year
  ▪ Radiographically using cone beam computed tomography: percent of change in periapical lesion size in cubic millimeters

SECONDARY OUTCOMES:
percent of change in root length | 1 year
  Radiographically using CBCT: percent of change in length in millimeters
percent of change in apical area | 1 year
  Radiographically using CBCT: percent of change in apical area in squared millimeters.
percent of change in root width | 1 year
  Radiographically using CBCT: percent of change in root width in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Future University in Egypt, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No